CLINICAL TRIAL: NCT05154227
Title: Health@NUS - Studying Health Behaviours and Well-being During the Student-to-Work Life Transition Using mHealth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Health Promotion Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Dr Falk Mueller-Riemenschneider, Associate Professor, National University of Singapore
Other Study IDs: Health@NUS
Record Dates: First submitted 2021-09-16; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: mhealth; young adults cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate body-weight and behavioural trajectories, as well as their underlying individual, social, and environmental determinants from University to early working life. The study employs mHealth approaches in the form of a smartphone app and smart wearables to collect health behaviour and related information to answer the following research questions:

1. To what extend do health behaviours (activity, diet, and sleep), body weight, and mental well-being change during the transition from university to early working life?
2. What is the relationship between health behaviours and mental well-being, and how does it differ at different stages of the transition from University to early working life?
3. What are the determinants of physical activity, healthy eating and sleep in university students and young working adults?
4. Do these determinants differ at different stages of the student to work life transition?
5. If so, how do these differences in these determinants relate to changes in health behaviours, weight status, and mental well-being?

DETAILED DESCRIPTION:
This is a prospective cohort study. The study period for each participant is 2 years. Participants are required to download the study's smartphone app and wear the assigned smartwatch to collect various information (including step counts and sleep time). Physical measurements are taken in person at baseline, 12 months and 24 months visits. These measurements include height, weight, waist circumference, resting heart rate and blood pressure.

Questionnaires administered at baseline, 12 months and 24 months include:

* Demographics (age, gender, religion, socio-economic status, education level)
* Personality
* Dietary intake and habits
* Physical activity, sedentary behavior and screen time
* Active and passive transport use
* Smoking habit
* Sleep quality
* Mental health and wellness
* Medical history
* Women's health-related

Participants will also receive occasional surveys sent to their smartphone through the study app. These surveys will include questions about sleep, diet, technology use, binge drinking, smoking, physical activities and/or emotions.

ELIGIBILITY:
Inclusion Criteria:

* Full time National University of Singapore students (undergraduate and postgraduate)
* Singapore Citizen or Permanent Resident;
* Has a Singapore registered mobile number• Owns a mobile phone with operating system that is compatible with the study app (iOS 10 or Android 7 and above);
* Able to make the upfront deposit of $20 and able to set up the Direct Debit Authorization (DDA) for possible deductions by HPB;
* Able to understand the study procedure during the informed consent taking process.

Exclusion Criteria:

* Students who will be overseas for more than 6 weeks per trip during the study period (e.g. involved in overseas exchange/internship programmes or stationed overseas) or travelling frequently;
* Students who are not able to set up the DDA via online method will be excluded;
* Students who has worked in a full-time position for more than a year previously;
* Pregnant women will be excluded only at the point of recruitment.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a cohort of National University of Singapore (NUS) (undergraduate and postgraduate) students.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Changes in health behaviours - physical activity | Baseline, 12 and 24 months follow up
Changes in health behaviours - dietary pattern | Baseline, 12 and 24 months follow up
Changes in health behaviours - sleep pattern | Baseline, 12 and 24 months follow up
Changes in health behaviours - mental well-being | Baseline, 12 and 24 months follow up

SECONDARY OUTCOMES:
Blood pressure (mmHG) | Baseline, 12 and 24 months follow-up
Resting heart rate (bpm) | Baseline, 12 and 24 months follow-up
Body Mass Index (kg/m^2) | Baseline, 12 and 24 months follow-up
Waist circumference (cm) | Baseline, 12 and 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Falk Müller-Riemenschneider, Principal Investigator — National University of Singapore
Locations (1):
- Saw Swee Hock School of Public Health, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng S, Chua XH, Edney SM, Goh CM, Tai BC, Chia J, Koek D, van Dam RM, Muller-Riemenschneider F. Movement and dietary behaviours and mental health among university students: the Health@NUS study. BMC Public Health. 2025 Sep 24;25(1):3100. doi: 10.1186/s12889-025-24340-5. PMID 40993637
- [Derived] Chua XH, Edney SM, Muller AM, Petrunoff NA, Whitton C, Tay Z, Goh CMJL, Chen B, Park SH, Rebello SA, Low A, Chia J, Koek D, Cheong K, van Dam RM, Muller-Riemenschneider F. Rationale, Design, and Baseline Characteristics of Participants in the Health@NUS mHealth Augmented Cohort Study Examining Student-to-Work Life Transition: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2024 Jul 17;13:e56749. doi: 10.2196/56749. PMID 39018103
- [Derived] Edney S, Goh CM, Chua XH, Low A, Chia J, S Koek D, Cheong K, van Dam R, Tan CS, Muller-Riemenschneider F. Evaluating the Effects of Rewards and Schedule Length on Response Rates to Ecological Momentary Assessment Surveys: Randomized Controlled Trials. J Med Internet Res. 2023 Oct 19;25:e45764. doi: 10.2196/45764. PMID 37856188